CLINICAL TRIAL: NCT03929913
Title: NHLBI DIR Transcatheter Mitral Cerclage Annuloplasty Early Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190088; 19-H-0088
Record Dates: First submitted 2019-04-26; First posted 2019-04-29 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Functional Mitral Regurgitation
Keywords: Ventricular Dysfunction; Functional Mitral Regurgitation; Heart Failure; Mitral Implant; Secondary Mitral Regurgitation
MeSH Terms: conditions — Ventricular Dysfunction; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcatheter Mitral Valve Cerclage Annuloplasty (Experimental): To evaluate the feasibility and safety of Transcatheter Mitral Cerclage Annuloplasty (TMCA) to treat symptomatic heart failure accompanied by mitral valve regurgitation despite optimal medical therapy.
  The TMCA implant is attached to a guidewire and pulled through the internal jugular sheath, along the coronary sinus, through the basal septum, through the tricuspid valve, and back out of the internal jugular sheath. The position of the TMCA implant is adjusted so that the coronary protection element lies directly over any underlying branch of the left coronary artery.
  Interventions: Device: Transmural Systems Transcatheter Mitral Cerclage Annuloplasty (TMCA)

INTERVENTIONS:
Device: Transmural Systems Transcatheter Mitral Cerclage Annuloplasty (TMCA) — The Transcatheter Mitral Cerclage Annuloplasty implant has two components, with or without a coronary artery protection element, and the wishbone lock with coronary sinus and right ventricular outflow track limbs. Procedure is performed from a trans-jugular venous approach. Coronary guidewires and microcatheters are used to navigate into a coronary vein to the target capture catheter. The implant is then attached to the back end of the guidewire and pulled out of the internal jugular sheath. The position of the implant is adjusted so the coronary protection element lies directly over any underlying branch of the left coronary artery. The wishbone lock is advanced over the two limbs of the implant and the desired tension is titrated to the degree of mitral regurgitation. Coronary angiography is performed to confirm there is no coronary compression. After desired tension has been achieved, the wishbone lock is locked and the two limbs of the implant are cut with a cutter catheter.

SUMMARY:
This research protocol tests a new technique and devices that we have developed to treat functional mitral valve regurgitation, called transcatheter mitral valve cerclage annuloplasty, otherwise known as "cerclage". Functional mitral valve regurgitation is a condition caused by damaged heart muscle involving the left ventricle which results in mitral valve leakage. This leakage causes heart failure (breathlessness and lack of energy especially when walking or exercising, and hospital admissions for fluid buildup).

This is an early feasibility study (EFS) evaluation of special devices, permanently implanted in the heart, to perform mitral cerclage annuloplasty. Mitral cerclage annuloplasty is a catheter procedure performed under X-ray and ultrasound guidance without surgery. The cerclage devices compress the mitral valve like a purse-string. The cerclage device has a special feature that prevents a coronary artery from getting squeezed as part of this purse-string.

The protocol has been changed to allow patients who have mitral valve regurgitation despite prior Mitra-Clip treatment, and to allow patients who have symptomatic heart failure with mild mitral regurgitation.

DETAILED DESCRIPTION:
Functional mitral regurgitation (also known as secondary mitral regurgitation) is a common complication of left ventricular dysfunction. Ventricular dysfunction leads to dilation, which in turn leads to mitral annular dilation and leaflet traction. This causes a failure of coaptation of the otherwise intact leaflets of the mitral valve, leading to regurgitation through a central orifice between the mal-coapting leaflet tips. Functional mitral regurgitation contributes to heart failure symptoms. Transcatheter Mitral Cerclage Annuloplasty (TMCA) is a new catheter technique that reduces the septal-lateral dimension of the dilated annulus through circumferential compression, prevents extrinsic compression and entrapment of coronary arteries by incorporating a protection element, and exhibits planar discordance that achieves annular reduction even when the coronary sinus is anatomically located along the posterior left atrial wall. This is an entirely right-sided procedure and device.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults age >=21 years
  2. Symptomatic functional mitral valve regurgitation

     1. Mild or greater mitral valve regurgitation, LVEF <= 0.50, and NYHA class III - IV heart failure
     2. Moderate or greater mitral valve regurgitation and NYHA II - IV heart failure, irrespective of LV systolic function
  3. On optimal medical therapy for at least one month
  4. Left ventricular ejection fraction >=0.20 assessed by echocardiography, CT, or CMR
  5. Suitable coronary venous anatomy for Transcatheter Mitral Cerclage Annuloplasty based on pre-procedural cardiac CT or coronary venogram
  6. Concordance of the Study Eligibility Committee
  7. If present, a MitraClip was implanted at least 30 days previously

EXCLUSION CRITERIA:

1. Subjects unable to consent to participate
2. Subjects unwilling to participate or unwilling to return for study follow-up activities.
3. Prior cardiac implanted electronic devices (CIED) likely to be entrapped by cerclage.

   -- Candidates with coronary sinus or left ventricular pacing or defibrillation leads that are not likely to be entrapped by cerclage, evident on baseline CT or angiogram, are eligible to participate.
4. TAVR within 6 weeks
5. Intended concurrent structural heart procedure, such as aortic or tricuspid valve intervention
6. Aortic stenosis more than mild in severity
7. Single-leaflet MitraClip detachment, if present
8. Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Carilion Medical Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The authors are willing to share de-identified subject data upon reasonable request.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-H-0088.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen subjects consented and underwent cerclage procedures between May 2019 and February 2021, despite COVID-19-related delays.
Period: Overall Study
Arm/Group | Transcatheter Mitral Valve Cerclage Annuloplasty
Started | 19
Completed | 12
Not Completed | 7
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Failed Procedure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Transcatheter Mitral Valve Cerclage Annuloplasty
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Heart failure with reduced ejection fraction (HFrEF) [Count of Participants; unit: Participants] | 12
Heart failure with preserved ejection fraction (HFpEF) [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is Technical Success
Description: The primary endpoint is Technical success. This endpoint is measured at exit from the catheterization laboratory. All of the following must be present:
  1. Alive
  2. Successful deployment and correct positioning of a single intended Transcatheter Mitral Cerclage Annuloplasty (TMCA). Repositioning and recapture of the device, if needed, is not classified as failure.
  3. Retrieval of the TMCA delivery system
  4. Absence of TMCA-related coronary artery compression and absence of additional procedure such as percutaneous coronary intervention (PCI) to relieve coronary artery compression.
  5. No additional unplanned or emergency surgery or re-intervention related to the TMCA or delivery system.
Time Frame: 1 minute following procedure discharge (Exit from the catheterization laboratory)
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Cerclage Annuloplasty
Number analyzed (Participants) | 19
Participants | 17

2. Secondary Outcome: The Secondary Endpoint is Procedural Success
Description: The secondary endpoint is Procedural success This endpoint is measured at 30 days. All of the following must be present:
  1. Technical success
  2. No Transcatheter Mitral Cerclage Annuloplasty (TMCA) device-related Serious Adverse Events, defined as VARC-2 life-threatening bleeding, major vascular or cardiac complications related to the TMCA requiring unplanned reintervention or surgery.
Time Frame: Day 30 post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Cerclage Annuloplasty
Number analyzed (Participants) | 19
Participants | 16

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse event recording starts on Day (0) of the Transcatheter Mitral Cerclage Annuloplasty procedure and continues through the 12 month Follow Up. Reporting of serious adverse events (SAE) and serious adverse device effects (SADE) will continue at annual visits thereafter to year 5. Once the subject's 30 day follow up is completed, only serious adverse events (SAE), serious adverse device effects (SADE), unanticipated device effects (UADE) and unanticipated problems (UP) will be reported.
Arm/Group | Transcatheter Mitral Valve Cerclage Annuloplasty
All-Cause Mortality (participants affected / at risk) | 5/19
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Mitral Valve Cerclage Annuloplasty (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (4)
Atrioventricular block complete (Cardiac disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiogenic Shock-post cardiac arrest (Cardiac disorders) | 1 (1)
Torsade de Pointes (Cardiac disorders) | 1 (1)
Cardiac Chest pain (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 7 (18)
Myocardial infarction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hemoperitoneum with suspected clot overlaying left anterior liver left lobe (Injury, poisoning and procedural complications) | 1 (1) — hemoperitoneum with suspected clot overlaying left anterior liver left lobe post cardiac compressions with cardiac arrest response.
Transaminitis-Shock liver post cardiac arrest-elevated liver enzymes; moderate ascites on US. (Injury, poisoning and procedural complications) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
COVID infection, hospitalized. Unvaccinated (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Sodium low (Investigations) | 1 (1)
Colon cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Mitral Valve Cerclage Annuloplasty (N=19)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 13 (13)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inflammatory Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Episode of PAF during procedure requiring cardioversion (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Cardiac disorders) | 19 (19)
Cardiac Chest pain (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 5 (5)
Heart failure (Cardiac disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 2 (2)
Cardiac troponin I increased (Investigations) | 19 (19)
Creatinine increased (Investigations) | 5 (5)
Ejection fraction decreased (Investigations) | 2 (2)
BNP elevated post procedure (Investigations) | 5 (5)
NT-BNP elevated post procedure (Investigations) | 4 (4)
Elevated PCWP-post procedure from baseline (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 8 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Generalized itching post procedure (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Compression of left anterior descending artery (Injury, poisoning and procedural complications) | 1 (1) — Aborted implantation of cerclage device RT device causing compression of left anterior descending artery
Air embolization (Injury, poisoning and procedural complications) | 1 (1)
Cerclage device created compression of the LAD during cinching of the device. (Injury, poisoning and procedural complications) | 1 (1)
Crimp failure after tension element successfully traversed myocardium (Injury, poisoning and procedural complications) | 1 (1) — Crimp failure after tension element successfully traversed myocardium, during withdrawal from Gore Sheath.
Cutter Device malfunction (Injury, poisoning and procedural complications) | 1 (1)
Throat pain and tongue swelling (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Adenocarcinoma of the right lower lobe lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other
A Publications Committee comprised of the NIH Principal Investigator (PI) and Investigators participating in the study, as appropriate, will be formed to oversee the publication and presentation of the study results, which will reflect the experience of all investigational sites. No publication or disclosure of study results will be permitted except under the terms and conditions of a separate written agreement between NIH PI and the non-NIH Investigator and/or the Investigator's institution.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT03929913/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03929913/ICF_001.pdf